CLINICAL TRIAL: NCT04715308
Title: Surgical and Patient-entered Experiences Following Urinary Reconstruction After Pelvic Exenteration for Locally Advanced and Recurrent Rectal Cancer
Brief Title: Patient Experiences Following Urinary Diversion as Part of Surgery for Advanced and Recurrent Rectal Cancer
Acronym: Pelvex 3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Des Winter, Professor Des C Winter, Consultant Gastronitestinal Surgeon, St Vincent's University Hospital, Ireland
Other Study IDs: STVINCENTSIRELAND
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Patient Satisfaction; Quality of Life; Patient Participation
Keywords: Rectal cancer; Locally advanced and recurrent rectal cancer; Advanced pelvic cancer; Urinary diversion for rectal cancer; Quality of life
MeSH Terms: conditions — Patient Satisfaction; Patient Participation; Rectal Neoplasms | interventions — Urinary Diversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Urinary diversion — The formation of a stoma to divert urine to the skin because of the need to resect the bladder as part of surgery for advanced pelvic malignancy

SUMMARY:
The outcomes of patients who undergo radical surgery for locally advanced and recurrent rectal cancer have improved vastly, but there is a lack of emphasis on the quality-of-life outcomes of these patients. This study will assess the patient experience of having a stoma for urinary diversion as part of surgery for advanced pelvic malignancy. This will be assessed at regular intervals both before and after surgery with the goal of increasing awareness of patient beliefs and concerns with regards to their stomas and to devise interventions that will improve their quality-of-life.

DETAILED DESCRIPTION:
Considerable progress has been made in the management of advanced and recurrent pelvic cancer over the last few decades. However, much emphasis has been placed on surgical and hospital-related outcomes. In recent years, there has been an increased focus on patient quality-of-life following major abdominopelvic surgery. However, there is a lack of updated evidence on how patients manage and perceive their stomas. Managing a stoma is a difficult task for patients and can adversely effect their quality-of-life. This study will investigate specifically the impact of managing a urostomy or ileal conduit. Patients will be contacted via an anonymized, opt-in SMS or email to answer a questionnaire, having previously been provided with a patient information leaflet. This will take approximately 5 minutes to complete and will be carried out just prior to and at 1, 3, 6, 9 and 12 months post-operatively. All of this data will be collated and published as part of a wider investigation in to patient quality-of-life following major abdominal and pelvic surgery. This study will be carried out in 35 countries.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven advanced rectal cancer
* Has undergone urinary diversion/reconstruction
* Aged 18 years or older
* Able and willing to give written, informed consent
* Able to access email/internet

Exclusion Criteria:

* Strong evidence of metastatic or peritoneal disease
* Palliative exenteration
* Non-rectal origin of primary tumour
* Colonic obstruction
* Inability to answer online questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients who are undergoing surgery for locally advanced or recurrent rectal cancer and are undergoing a urinary diversion or reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
To determine the 30-day complication rate of urinary diversion/reconstruction following pelvic exenteration | 2 years
  Morbidity of urinary diversion/reconstruction
To assess the impact of urinary diversion/reconstruction subtypes on quality-of-life | Before surgery and at 1, 3, 6, 9 and 12 months respectively
  Patient-reported outcomes assessing their quality-of-life

SECONDARY OUTCOMES:
To assess the longer-term complications associated with urinary diversion/reconstruction | 1 month - 12 months
  Morbidity of urinary diversion or reconstruction over longer than 1 month but less than 1 year
To measure the rate of reintervention for complications associated with urinary diversion/reconstruction | 12 months
  Rate of reintervention

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
No individual patient date other than their responses to the questionnaire will be collected or shared.